CLINICAL TRIAL: NCT07155395
Title: Relationship Between Inflammatory and Hematological Indices and Coronary Artery Disease Severity and Outcome Among Diabetic Patients Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Inflammatory and Hematological Indices in Diabetic STEMI Patients Undergoing Primary PCI
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, David Emil Efraim Danial, Resident Cardiologist, Assiut University
Other Study IDs: Markers in Diabetic STEMI
Record Dates: First submitted 2025-08-24; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: STEMI; Diabete Mellitus
Keywords: STEMI; Diabetes; No reflow; SYNTAX; Hb/RDW; RDW/PDW; NAR; SIRI; SII; CRP; PPCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic STEMI Patients: Patients presenting with ST-segment elevation myocardial infarction (STEMI) and a confirmed diagnosis of diabetes mellitus, undergoing primary percutaneous coronary intervention (PCI).
- Non-Diabetic STEMI Patients: Patients presenting with STEMI and no history or diagnosis of diabetes, undergoing primary PCI.

SUMMARY:
ST-segment Elevation Myocardial Infarction (STEMI) remains a major cause of mortality despite the adoption of Primary Percutaneous Coronary Intervention (PPCI) as the standard treatment. However, outcomes still vary significantly among patients, especially between diabetic and non-diabetic cohorts.

The research question driving this study is: Can hematologic, inflammatory, and thrombotic indices serve as reliable prognostic tools in predicting the no-reflow phenomenon and coronary artery disease (CAD) severity in STEMI patients, particularly among those with diabetes mellitus?

Recent literature identifies inflammation as a key contributor to the pathogenesis and outcomes of Acute Coronary Syndrome (ACS), including the no-reflow phenomenon and Major Adverse Cardiovascular Events (MACE). Markers such as C-reactive protein (CRP), Neutrophil-to-Albumin Ratio (NAR), Red Cell Distribution Width (RDW), Platelet Distribution Width (PDW), Hemoglobin-to-Red Cell Distribution Width ratio (Hb/RDW), and the RDW/PDW ratio have shown individual correlations with poor outcomes. Emerging indices such as the Systemic Immune-Inflammation Index (SII) and the Systemic Inflammatory Response Index (SIRI) further integrate immune and inflammatory components and have shown promise in early risk stratification.

The current strategy in many cardiac centers relies on angiographic and clinical indicators, which may be insufficient for individualized risk prediction. Hence, incorporating accessible and cost-effective blood-based markers could significantly enhance prognostic accuracy.

The rationale of this research lies in comparing these indices in diabetic versus non-diabetic STEMI patients, aiming to stratify risk, predict no-reflow, assess coronary artery disease burden using the SYNTAX score, and identify those at risk for early adverse outcomes.

DETAILED DESCRIPTION:
ST-segment Elevation Myocardial Infarction (STEMI) is a critical form of Acute Coronary Syndrome (ACS), resulting from abrupt plaque rupture and thrombotic coronary occlusion. Despite the widespread application of Primary Percutaneous Coronary Intervention (PPCI), STEMI remains one of the leading causes of mortality. Therefore, early stratification and prediction of outcomes is essential.

Recent evidence highlights that, in addition to thrombosis, inflammation plays a crucial role in the pathophysiology of ACS. This has prompted increasing interest in novel inflammatory and hematological biomarkers as promising prognostic tools. These indices are simple, cost-effective, and clinically relevant for outcome prediction.

The markers evaluated in this study include both inflammatory indices (e.g., C-reactive protein [CRP], Neutrophil-to-Albumin Ratio [NAR]) and thrombotic/hematological indices (e.g., Red Cell Distribution Width [RDW], Platelet Distribution Width [PDW], Hemoglobin-to-Red Cell Distribution Width ratio [Hb/RDW], and RDW/PDW ratio). Some of these have already been established as strong predictors of adverse outcomes in STEMI patients, while others remain under investigation. Moreover, their differential prognostic value in diabetic versus non-diabetic STEMI populations remains an area of ongoing research.

Among the markers for inflammation, C-reactive protein (CRP) has been shown to be strongly associated with increased in-hospital mortality among STEMI patients. Another important marker is the Neutrophil-to-Albumin Ratio (NAR), which combines indicators of systemic inflammation and nutritional status. Higher NAR levels have been linked with poor in-hospital outcomes in STEMI.

This study also evaluates hematological and thrombotic indices. Red Cell Distribution Width (RDW), an indicator of anisocytosis, is a well-studied parameter. Increased RDW levels have been associated with worse outcomes in cardiovascular diseases (CVD) and heart failure. Platelet Distribution Width (PDW)-a marker of platelet activation and heterogeneity-has been identified as a strong independent predictor of the no-reflow phenomenon. An elevated RDW/PDW ratio is thought to represent systemic stress and a prothrombotic state, making it a compelling predictor of poor clinical and angiographic outcomes such as no-reflow.

The Hemoglobin-to-Red Cell Distribution Width ratio (Hb/RDW) is a novel indicator. A lower Hb/RDW ratio reflects reduced tissue oxygenation and erythropoietic dysfunction, both of which are linked to poor myocardial recovery, no-reflow, and higher SYNTAX scores.

The no-reflow phenomenon, which these markers help anticipate, is defined as inadequate myocardial perfusion through a segment of the coronary circulation in the absence of mechanical obstruction.

In addition to traditional markers, the Systemic Immune-Inflammation Index (SII) and the Systemic Inflammatory Response Index (SIRI) have recently gained attention. Both are calculated using peripheral blood counts and provide insight into the interplay between inflammation, thrombosis, and immune regulation:

Systemic Immune-Inflammation Index (SII): Platelet count × Neutrophil count / Lymphocyte count.

This index combines neutrophil-driven inflammation, platelet-related thrombosis, and lymphocyte-mediated immune regulation. SII has been recognized as a powerful predictor of no-reflow, MACE, and mortality in cardiovascular patients.

Systemic Inflammatory Response Index (SIRI): Monocyte count × Neutrophil count / Lymphocyte count.

This index reflects systemic inflammation and monocyte activity in atherosclerosis. Elevated SIRI has been associated with higher SYNTAX scores, no-reflow, and adverse cardiovascular outcomes.

Thus, exploring the association between different hematologic-inflammatory indices-including Hb/RDW, RDW/PDW, NAR, SII, SIRI, Neutrophil-to-Lymphocyte Ratio (NLR), and Platelet-to-Lymphocyte Ratio (PLR)-with no-reflow, coronary artery disease severity, and short-term outcomes in diabetic versus non-diabetic STEMI patients undergoing PPCI remains clinically relevant and needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Assiut University cardiac catheterization laboratory with ST-segment Elevation Myocardial Infarction (STEMI).
* Managed with primary percutaneous coronary intervention (PPCI).

Exclusion Criteria:

* Patients not eligible for PPCI.
* Patients who underwent thrombolytic therapy or received anti-thrombotics prior to hospital arrival.
* Prior coronary intervention: history of PCI or CABG.
* Known hematological disorders:

Thalassemia (microcytic anemia, normal iron profile, HbA2 ≥ 3.5% or elevated HbF).

Myelodysplastic syndromes (unexplained cytopenias with ≥10% dysplasia in bone marrow aspirate).

Leukemia (persistent leukocytosis or pancytopenia, blasts ≥20% in peripheral blood).

* Active infection or sepsis at admission (e.g., fever, leukocytosis, elevated CRP <100 mg/L without cardiac cause).
* Known autoimmune or chronic inflammatory diseases (e.g., systemic lupus erythematosus).
* Known or newly diagnosed malignancy.
* End-stage renal disease (eGFR <30 ml/min/1.73 m² or on dialysis).
* Advanced hepatic impairment (Child-Pugh class C; bilirubin >3 mg/dL or ALT/AST >3× upper limit of normal).
* Recent blood transfusion within 3 months.
* Recent use of steroids, chemotherapy, or immunosuppressive drugs.
* Mechanical complications or cardiogenic shock prior to or during STEMI presentation (e.g., papillary muscle rupture, ventricular septal defect, need for intra-aortic balloon pump).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients present with STEMI and undergoing primary percutaneous coronary intervention in Assiut university heart hospital (AUHH). Patients will be categorized into 2 groups: Diabetics and non-diabetics based on HbA1c.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | Peri-procedural
  Composite outcome including heart failure, fatal arrhythmia, death, re-infarction, stroke, and urgent target vessel revascularization. The prognostic value of various biomarkers (Hb/RDW, RDW/PDW, NAR, SII, SIRI) will be assessed in diabetic vs. non-diabetic STEMI patients during admission.
Angiographic outcomes including No Reflow Phenomenon | At time of Primary PCI (within 24 hours of admission)
  Assessment of angiographic outcomes following primary percutaneous coronary intervention (PPCI), with a specific focus on the incidence of the no-reflow phenomenon. No-reflow will be defined as inadequate myocardial perfusion in the absence of mechanical obstruction.

SECONDARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | Up to 6 months post-PCI
  Composite outcome including heart failure, fatal arrhythmia, death, re-infarction, stroke, and urgent target vessel revascularization. The prognostic value of various biomarkers (Hb/RDW, RDW/PDW, NAR, SII, SIRI) will be assessed in diabetic vs. non-diabetic STEMI patients over the 6-month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelghany, Study Director — Assiut University; Heba Mahmoud Elnaggar, Study Director — Assiut University

REFERENCES:
- [Background] Li H, Xu Y. Association between red blood cell distribution width-to-albumin ratio and prognosis of patients with acute myocardial infarction. BMC Cardiovasc Disord. 2023 Feb 3;23(1):66. doi: 10.1186/s12872-023-03094-1. PMID 36737704
- [Background] Milano et al., 2019 (CRP predictor in STEMI; Int J Cardiovasc Sci)
- [Background] Kılıç et al., 2024 (Hb/RDW ratio in ACS)
- [Background] Cui H, Ding X, Li W, Chen H, Li H. The Neutrophil Percentage to Albumin Ratio as a New Predictor of In-Hospital Mortality in Patients with ST-Segment Elevation Myocardial Infarction. Med Sci Monit. 2019 Oct 19;25:7845-7852. doi: 10.12659/MSM.917987. PMID 31628741
- [Background] Sahinkus S, Cakar M, Yaylaci S, Aydin E, Can Y, Kocayigit I, Osken A, Akdemir R, Gunduz H. HEMATOLOGICAL MARKERS OF THE NO-REFLOW PHENOMEN ON IN-PATIENTS UNDERGOING PRIMARY PERCUTANEOUS CORONARY INTERVENTION. Georgian Med News. 2016 May;(254):26-32. PMID 27348163
- [Background] Milwidsky A, Ziv-Baran T, Letourneau-Shesaf S, Keren G, Taieb P, Berliner S, Shacham Y. CRP velocity and short-term mortality in ST segment elevation myocardial infarction. Biomarkers. 2017 May-Jun;22(3-4):383-386. doi: 10.1080/1354750X.2017.1279218. Epub 2017 Jan 25. PMID 28055283
- [Background] Bao D, Luo G, Kan F, Wang X, Luo J, Jiang C. Prognostic value of red cell distribution width in patients undergoing percutaneous coronary intervention: a meta-analysis. BMJ Open. 2020 Sep 10;10(9):e033378. doi: 10.1136/bmjopen-2019-033378. PMID 32912972
- [Background] Babes EE, Zaha DC, Tit DM, Nechifor AC, Bungau S, Andronie-Cioara FL, Behl T, Stoicescu M, Munteanu MA, Rus M, Toma MM, Brisc C. Value of Hematological and Coagulation Parameters as Prognostic Factors in Acute Coronary Syndromes. Diagnostics (Basel). 2021 May 9;11(5):850. doi: 10.3390/diagnostics11050850. PMID 34065132